CLINICAL TRIAL: NCT05248763
Title: Taiwan Cancer Moonshot Project: 1. Next-generation Pathway of Taiwan Cancer Precision Medicine (Subjective Aim 1- Taiwan Cancer Moonshot Project); 2. Development of Novel Treatments for Major Diseases (Subproject 5 - Multiomic Big Data-based Intelligent Navigation System for Precision Oncology)
Brief Title: Taiwan Cancer Moonshot Project
Status: Recruiting | Type: Observational
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AS-IRB-BM-17056
Record Dates: First submitted 2022-01-24; First posted 2022-02-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Malignant Neoplasm of Body of Stomach in Situ
Keywords: lung cancer; breast cancer; gastric cancer; pancreatic cancer; ovarian cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to establish multiomic big data under strictly collected clinical samples from tumors, adjacent normal tissue, blood, and clinical data then analyze by using integrated proteomics and genetics platform.

DETAILED DESCRIPTION:
Multiomic integrative analysis is an effective strategy to facilitate the investigation of molecular mechanism, cause, and early intervention of specific diseases. Gastric cancer is specifically chosen for our research target to decrease its incidence and improve survival. To increase precision diagnosis, prognosis and precision therapy, patients from Taiwan are selected as cohort subjects. The aim of this study is to establish multiomic big data under strictly collected clinical samples from tumors, adjacent normal tissue, blood, and clinical data then analyze by using integrated proteomics and genetics platform. Genome, transcriptome, genomic methylation, proteomics, and post-translational modification will be used to construct a map for determine the in-depth carcinogenesis of gastric cancer and strategies for cancer early diagnosis, prevention, and targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer, breast cancer, gastric cancer, pancreatic cancer, ovarian cancer

Exclusion Criteria:

* other cancer types

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: lung cancer, breast cancer, gastric cancer, pancreatic cancer, ovarian cancer in Taiwan
Sampling Method: Probability Sample
Enrollment: 4190 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Collected clinical samples from tumors, adjacent normal tissue, blood, and clinical data | Through study completion, an average of 2 to 3 year
  Analyze collected clinical samples by using integrated proteomics and genetics platform (genome, transcriptome, genomic methylation, proteomics, and post-translational modification)

SECONDARY OUTCOMES:
Differential expressed genes and proteins in tumor | Through study completion, an average of 4 year
  The relative difference, or fold change of expressed genes and proteins (tumors vs adjacent normal tissue)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ju Chen, PhD, Study Director — Distinguished Research Fellow
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan